CLINICAL TRIAL: NCT03511066
Title: A Phase IIb, Randomized, Double-blind, Multicenter, Placebo-controlled Study Evaluating the Efficacy and Safety of CT-P27 in Subjects With Acute Uncomplicated Influenza A Infection
Brief Title: A Study to Evaluate the Efficacy and Safety of CT-P27 in Acute Uncomplicated Influenza A Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: CT-P27 2.2 is inactivated
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P27 2.2
Record Dates: First submitted 2018-02-28; First posted 2018-04-27 (Actual); Results first posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-08

CONDITIONS: Influenza A
Keywords: efficacy; safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CT-P27 90 mg/kg (Experimental): CT-P27 will be administrated once in IV infusion.
  Interventions: Drug: CT-P27 90 mg/kg
- CT-P27 45mg/kg (Experimental): CT-P27 will be administrated once in IV infusion.
  Interventions: Drug: CT-P27 45 mg/kg
- Placebo (Placebo Comparator): Placebo will be administrated once in IV infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CT-P27 90 mg/kg — Influenza A treatment drug.
  Other Names: CT-P27
  Arms: CT-P27 90 mg/kg
Drug: CT-P27 45 mg/kg — Influenza A treatment drug.
  Other Names: CT-P27
  Arms: CT-P27 45mg/kg
Drug: Placebo — Placebo.
  Arms: Placebo

SUMMARY:
This study is a Phase IIb, Randomized, Double-blind, Multicenter, Placebo-controlled study evaluating the efficacy and safety of CT-P27 in subjects with acute uncomplicated influenza A infection.

DETAILED DESCRIPTION:
This study is a Phase IIb, Randomized, Double-blind, Multicenter, Placebo-controlled study. All enrolled subjects will be given a single dose of 90 mg/kg CT-P27, 45 mg/kg CT-P27, or placebo intravenously over 90 minutes (±15 minutes) on Day 1 and then followed by Day 110.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects between the ages of 19 and 64 years, both inclusive
* Diagnosed with influenza A at screening using rapid influenza diagnostic test
* Onset of influenza symptoms and fever is within 48 hours at screening
* At least 2 of symptoms (moderate to severe in intensity)
* ≥38.0'C body temperature at screening

Exclusion Criteria:

* Taking antiviral treatment for influenza or has a history of using these antivirals within 14 days prior to the administration of study drug
* Positive influenza B or A+B infection

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MoonSun Choi, Study Director — Celltrion Inc.
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo will be administrated once in IV infusion.
  Placebos: Placebo.
Period: Overall Study
Arm/Group | CT-P27 90 mg/kg | CT-P27 45mg/kg | Placebo
Started | 88 | 90 | 50
Completed | 85 | 85 | 47
Not Completed | 3 | 5 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 3
Not completed — Lost to Follow-up | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P27 90 mg/kg | CT-P27 45mg/kg | Placebo | Total
Number analyzed (Participants) | 88 | 90 | 50 | 228
Age, Continuous [Median (Full Range); unit: years] | 38.5 [19 to 63] | 40.0 [19 to 64] | 34.5 [19 to 60] | 38.0 [19 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 26 | 112
  Male | 45 | 47 | 24 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 88 | 90 | 50 | 228
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 88 | 90 | 50 | 228
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 88 | 90 | 50 | 228
Positive rapid influenza diagnostic test at screening [Count of Participants; unit: Participants] | 88 | 89 | 50 | 227
Influenza A confirmation [Count of Participants; unit: Participants]
  by cell culture or qPCR | 87 | 86 | 48 | 221
  Not detected | 1 | 4 | 2 | 7
Influenza A subtype [Count of Participants; unit: Participants]
  Influenza A/H1 | 5 | 2 | 4 | 11
  Influenza A/H3 | 82 | 83 | 44 | 209
  Unknown | 0 | 1 | 0 | 1
  Not applicable | 1 | 4 | 2 | 7
Total influenza symptom score at screening [Mean (Full Range); unit: Averaged for each symptoms' score] — Average score of symptoms (Cough, Sore throat, Headache, Nasal congestion, Feeling feverish, Body aches and pains, Fatigue [Tiredness], Neck pain, Interrupted sleep and Loss of appetite) by Influenza Intensity and Impact Questionnaire (FluiiQ™): 0=None, 1=Mild, 2=Moderate, 3=Severe
  Averaged for each symptoms' score | 2.08 [1.0 to 3.0] | 2.05 [0.8 to 3.0] | 2.12 [0.8 to 3.0] | 2.08 [0.8 to 3.0]
Body temperature at screening [Mean (Standard Deviation); unit: °C] | 38.1 (0.74) | 38.3 (0.81) | 38.1 (0.65) | 38.2 (0.75)

OUTCOME MEASURES:

1. Primary Outcome: Time to Resolution of Influenza Symptoms and Fever
Description: Time to resolution of influenza symptoms (cough, sore throat, nasal congestion, headache, feeling feverish, body aches and pains, and fatigue) and fever (<37.8)
Time Frame: Twice a day (Morning and Evening) from Day 1 to Day 8
Population: The intent-to-treat-infected (ITTI) population defined as all randomized subjects with confirmed influenza A by quantitative polymerase chain reaction (qPCR) or cell culture.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CT-P27 90 mg/kg | CT-P27 45mg/kg | Placebo
Number analyzed (Participants) | 87 | 86 | 48
Days | 3.74 [2.72 to 4.46] | 3.69 [2.81 to 4.25] | 5.72 [3.65 to NA] — The upper limit of 95% CI was not calculated due to insufficient number of participants with events (resolution of influenza symptoms and fever).

ADVERSE EVENTS:
Time Frame: up to Day 110/end-of-study (EOS) visit
Arm/Group | CT-P27 90 mg/kg | CT-P27 45mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/90 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/88 | 5/90 | 1/50
Other Adverse Events (participants affected / at risk) | 8/88 | 8/90 | 6/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P27 90 mg/kg (N=88) | CT-P27 45mg/kg (N=90) | Placebo (N=50)
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P27 90 mg/kg (N=88) | CT-P27 45mg/kg (N=90) | Placebo (N=50)
Diarrhoea (Gastrointestinal disorders) | 3 | 7 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 2 | 1

LIMITATIONS AND CAVEATS:
All death, 'treatment-emergent' serious adverse events and 'treatment-emergent' adverse events were summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT03511066/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT03511066/SAP_001.pdf